CLINICAL TRIAL: NCT04616898
Title: Analysis of the Performance of 1060 nm Diode Laser and Radiofrequency Intended for Fat Reduction Prior to Abdominoplasty
Brief Title: Analysis of the Performance of 1060 nm Diode and Radio Frequency Prior to Abdominoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Venus Concept (Industry)
Collaborators: University of Texas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BL0519; STU2019-1160 (Other: UTSW)
Record Dates: First submitted 2020-07-21; First posted 2020-11-05 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Adipose Tissue Atrophy
Keywords: Adipose; Fat
MeSH Terms: conditions — Platelet Glycoprotein IV Deficiency

STUDY DESIGN:
Intervention Model Description: For this study, there will be three treatment groups in total. Details of each treatment are depicted in the addendum below. Groups 1 (laser only- 6 visits) and 2 (laser plus radiofrequency- 4 visits) will each consist of one patient. Group 3 (multiple vs. single laser treatments - 5 visits) will consist of three patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Diode Laser Treatment Only (Active Comparator): Group 1: Patient 1- Laser Only This patient will present 20+, 14, 7, and 1 days prior to his/her scheduled abdominoplasty. Between 20 and 30 days prior, the patient will receive the first laser treatment on the 20+ day site 1. 14 days prior, the patient will receive laser treatment on the 14 day site 2. 7 days prior, the patient will receive laser treatment on the 7 day site 3. 1 day prior to the scheduled abdominoplasty, the patient will receive laser treatment on the 24 hour site 4.
  Interventions: Device: Venus Bliss
- Diode Laser and RadioFrequency Treatment (Active Comparator): This patient will present 14 days and 7 days prior to his/her scheduled abdominoplasty. 14 days prior, the patient will be treated at site 1 with the laser and radiofrequency and site 3 with the laser only. 7 days prior, the patient will be treated at site 2 with the laser and radiofrequency and site 4 with the laser only.
  Interventions: Device: Venus Bliss
- Multiple Diode Treatments (Active Comparator): These patients will present for three treatments, each four weeks apart, with the abdominoplasty scheduled four weeks following the last laser treatment. These patients will receive laser treatment every four weeks for twelve weeks on the sites labelled Multiple Tx below (sites 1 and 2) on Days -90, -60, and -30 prior to abdominoplasty. At the final treatment (Day -30), two additional diodes will be placed on the sites labelled Single Tx below (sites 3 and 4). 4 diodes total will be used at this visit. Four weeks following this last treatment, the scheduled abdominoplasty will be performed and the pannus containing the treated tissue will be excised.
  Interventions: Device: Venus Bliss

INTERVENTIONS:
Device: Venus Bliss — The Venus Bliss™ system is an aesthetic medical device designed to non-invasively reduce subcutaneous adipose tissue of the abdominal area and flanks. It is intended for use in individuals with a Body Mass Index (BMI) of 30 or less. The device consists of an external treatment component and an internal control component. The treatment console is a 1060nm diode laser applicator and a radio frequency applicator. In addition, a Bliss Belt is provided with the system to properly secure one or more applicators to the patient's body during treatment. Finally, the touchscreen monitor is used by the clinician to control the setting display on the main console. It also keeps the clinician informed of the device's status and operating parameters.

SUMMARY:
To evaluate the safety and efficacy of treatment with 1060nm diode laser and radio frequency to be analyzed through histological and molecular analysis.

DETAILED DESCRIPTION:
The Primary Objectives of this protocol are to evaluate the safety and efficacy of treatment with 1060nm diode laser and radio frequency for use in aesthetic dermatological procedures requiring the ablation, excision, incision, or coagulation of soft tissue. Efficacy will be analyzed through histological and molecular analysis. Safety will be analyzed by monitoring the occurrence of any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are currently seeking abdominoplasty surgery and are consenting to their tissue that is being excised, to be tested
* Informed consent agreement signed by the subject.
* Fitzpatrick skin type I-V (Although the systems are cleared for all skin types I-VI, it is recommended to use the Matrix applicators on skin types I-V).
* Willingness to follow the treatment and follow-up schedule and the post-treatment care.
* For female candidates - post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study (i.e., oral contraceptives, IUD, contraceptive implant, barrier methods with spermicide, or abstinence).

Exclusion Criteria:

* Pregnant and/or breastfeeding.
* Having a history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treated area, unless treatment is conducted following a prophylactic regimen.
* Use of non-steroidal anti-inflammatory drugs (NSAIDS, e.g., ibuprofen-containing agents) one week before and after the treatment session.
* Use of retinoids, antioxidants or therapeutic skin nourishing supplements at medicinal concentration within 2 months of treatment or during the study and oral retinoids within 6 months of the study.
* Having received treatment with light, RF or other devices in the treated area within 6 months of treatment or during the study.
* Having received collagen/fat injections or other methods of augmentation with injected or implanted material in the treated area within 9 months of treatment or during the study.
* Having received Botox in the treated area within 6 months of treatment or during the study.
* Having undergone any other surgery in the treated area within 6 months of treatment (or more if skin has not healed completely) or during the study.
* History of keloid scarring or of abnormal wound healing.
* Suffering from current or history of significant skin conditions in the treated area or inflammatory skin conditions, including, but not limited to: active acne, excessive skin dryness, psoriasis, eczema, rash, rosacea (particularly severe open wound stage), varicella scars, open lacerations or abrasions and active cold sores or herpes sores prior to treatment (duration of resolution as per the Investigator's discretion) or during the treatment course.
* History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications.
* History of epidermal or dermal disorders (particularly if involving collagen or microvascularity).
* History of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation.
* Suffering from hormonal imbalance, as per the Investigator's discretion.
* Having a known anticoagulative or thromboembolic condition or taking anticoagulation medications one week prior to and during the treatment course (to allow inclusion, temporary cessation of use as per the subject's physician discretion).
* Having or undergoing any form of treatment for active cancer, or having a history of skin cancer or any other cancer in the areas to be treated, including actinic keratosis, presence of malignant or pre-malignant pigmented lesions.
* Suffering from significant concurrent illness, such as cardiac disorders, diabetes (type I or II), or pertinent neurological disorders.
* Vascular lesion, tattoo or permanent make-up in the treated area.
* Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study.
* Participation in a study of another device or drug within three month prior to enrollment or during the study.
* As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Changes in elastin as determined by histology on biopsied tissues | Day 1, Day 7, Day 14, Day 20-30 post-treatment
  Relative changes in protein abundance of biopsy samples taken post treatment compared to control or untreated group will be quantified using an image processing software based on fluorescence signal intensity. The change from baseline is calculated at each time frame.
Changes in collagen as determined by histology on biopsied tissues | Day 1, Day 7, Day 14, Day 20-30 post-treatment
  Relative changes in protein abundance of biopsy samples taken post treatment compared to control or untreated group will be quantified using an image processing software based on fluorescence signal intensity. The change from baseline is calculated at each time frame.
Changes in hyaluronic acid as determined by histology on biopsied tissues | Day 1, Day 7, Day 14, Day 20-30 post-treatment
  Relative changes in protein abundance of biopsy samples taken post treatment compared to control or untreated group will be quantified using an image processing software based on fluorescence signal intensity. The change from baseline is calculated at each time frame.

SECONDARY OUTCOMES:
Changes in elastin as a result of treatment measured by quantification of gene expression | Day 1, Day 7, Day 14, Day 20-30 post-treatment
  Biopsies of the treated tissue will be taken prior to treatment and post-treatment for gene expression analysis. This analysis will identify gene expression related to collagen formation and increased cell turnover.
Changes in collagen as a result of treatment measured by quantification of gene expression | Day 1, Day 7, Day 14, Day 20-30 post-treatment
  Biopsies of the treated tissue will be taken prior to treatment and post-treatment for gene expression analysis. This analysis will identify gene expression related to collagen formation and increased cell turnover.
Changes in hyaluronic acid as a result of treatment measured by quantification of gene expression | Day 1, Day 7, Day 14, Day 20-30 post-treatment
  Biopsies of the treated tissue will be taken prior to treatment and post-treatment for gene expression analysis. This analysis will identify gene expression related to collagen formation and increased cell turnover.
Quantification of the immune response following treatment | Day 1, Day 7, Day 14, Day 20-30 post-treatment
  Biopsies of the treated tissue will be taken prior to treatment and post-treatment for gene expression analysis. This analysis will identify gene expression related to the immune response.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Kenkel, MD, Principal Investigator — University of Texas
Locations (2):
- United States (2):
  - Dr. Brian Kinney Plastic Surgeon, Beverly Hills, California
  - University of Texas Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No